CLINICAL TRIAL: NCT01169025
Title: Fentanyl vs. Low-Dose Ketamine for the Relief of Moderate to Severe Pain in Aeromedical Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB_00040229
Record Dates: First submitted 2010-07-07; First posted 2010-07-23 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-06

CONDITIONS: Trauma; Pain
Keywords: Analgesia; Pain
MeSH Terms: conditions — Wounds and Injuries; Pain; Agnosia | interventions — Ketamine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Experimental): Subjects receive 0.3 mg/kg IV ketamine over 5 minutes and are evaluated every 10 minutes. Residual or recurring pain will be treated as needed with adjunctive open-label bolus dosing of IV fentanyl (1 mcg/kg) followed by repeat boluses as needed every 10 minutes during the flight. For this open-label portion of the flight, subjects are asked if they need additional pain medication every 10 minutes, unless an earlier, spontaneous request is made by the subject or the provider determines that more is needed. For the potential of rare ketamine side effects (dysphoria, anxiety, or agitation), 2 mg IV midazolam is given every 5 minutes as needed for any of these symptoms. Vital signs are measured continuously throughout the protocol. Blood pressure is measured at 5 minute intervals.
  Interventions: Drug: Ketamine
- Fentanyl (Active Comparator): Subjects receive 1 mcg/kg IV fentanyl over 5 minutes. After first dose administration, subjects are evaluated every 10 minutes. Residual or recurring pain is treated as needed with adjunctive open-label bolus dosing of IV fentanyl (1 mcg/kg) followed by repeat boluses as needed every 10 minutes during the flight. For this open-label portion of the flight, flight nurses will query participants regarding their desire for additional pain medication every 10 minutes unless an earlier, spontaneous request is made by the participant or the provider determines that more is needed. Vital signs are measured continuously throughout the protocol. Blood pressure is measured at 5 minute intervals.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Ketamine — Subjects receive 0.3 mg/kg IV ketamine over 5 minutes and are evaluated every 10 minutes. Residual or recurring pain will be treated as needed with adjunctive open-label bolus dosing of IV fentanyl (1 mcg/kg) followed by repeat boluses as needed every 10 minutes during the flight. For this open-label portion of the flight, subjects are asked if they need additional pain medication every 10 minutes, unless an earlier, spontaneous request is made by the subject or the provider determines that more is needed. For the potential of rare ketamine side effects (dysphoria, anxiety, or agitation), 2 mg IV midazolam is given every 5 minutes as needed for any of these symptoms. Vital signs are measured continuously throughout the protocol. Blood pressure is measured at 5 minute intervals.
  Other Names: Ketalar; Ketamine hydrochloride
  Arms: Ketamine
Drug: Fentanyl — Subjects receive 1 mcg/kg IV fentanyl over 5 minutes. After first dose administration, subjects are evaluated every 10 minutes. Residual or recurring pain is treated as needed with adjunctive open-label bolus dosing of IV fentanyl (1 mcg/kg) followed by repeat boluses as needed every 10 minutes during the flight. For this open-label portion of the flight, flight nurses will query participants regarding their desire for additional pain medication every 10 minutes unless an earlier, spontaneous request is made by the participant or the provider determines that more is needed. Vital signs are measured continuously throughout the protocol. Blood pressure is measured at 5 minute intervals.
  Other Names: Fentanil; Sublimaze; Actiq; Durogesic; Duragesic; Fentora; Onsolis; Instanyl
  Arms: Fentanyl

SUMMARY:
Often, patients transported by aeromedical systems do not receive enough medication to control and relieve their pain. The purpose of this study is to determine if pain treatment with intravenous (IV) ketamine is a better way to treat aeromedical patients' pain than the current treatment practices.

DETAILED DESCRIPTION:
Specific Aims: The aim of this study is to determine the efficacy, side effects and safety of sub-dissociative doses of ketamine in controlling acute traumatic pain in patients transported by an aeromedical system when compared to standard doses of fentanyl.

Research Hypothesis: Aeromedical transport patients with acute pain treated with intravenous ketamine show a clinically significant difference in mean numeric rating scale (NRS) pain scores as compared to those treated with fentanyl and show no increase in adverse events.

Background and Significance: Treatment of acute pain in aeromedical transport patients is important. Treatment may be limited by real or perceived concerns regarding analgesic side effects including sedation, loss of airway maintenance, and negative hemodynamic consequences. Ketamine used in sub-dissociative doses has strong analgesic properties while maintaining protective airway reflexes and demonstrating minimal adverse hemodynamic effects. It has been suggested as an ideal pre-hospital analgesic. Current literature regarding its use in the pre-hospital environment is limited.

Experimental Design: This prospective, double-blind, randomized trial compares 0.3 mg/kg of intravenous (IV) ketamine to 1 mcg/kg of IV fentanyl in adult aeromedical transport patients who require pain control. The primary outcome measure will be the change in NRS pain scores at ten minutes compared between the two groups. Secondary endpoints will include rates of adverse events, differences in the slope of NRS scores over time, the total amount of fentanyl/kg body weight/minute of flight required, overall research participant satisfaction with their level of pain relief at the end of the flight, and the subjective ranking of pain recall in comparison to other aspects of the patient's overall episode of care (pre-hospital, emergency department, inpatient, and post-discharge care), as measured at 30 days.

Data Analysis: Categorical variables will be analyzed using chi-square and Fisher's exact test. Means of normally distributed variables will be compared using Student's t-test, and distributions of non-normally distributed variables will be compared using Mann-Whitney U. Bayesian generalized linear mixed modeling will be employed to model the time-dependent change in NRS scores between intervention groups while accounting for the autocorrelation inherent in a repeated measures design. SAS statistical software (SAS v. 9.2, Cary, NC) and WinBUGS software will be used for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Moderate to severe acute, traumatic pain (self-reported NRS > 5)
* Ability to provide informed consent in English
* Flight destination to University of Utah Medical Center

Exclusion Criteria:

* Inability to use the NRS pain rating scale
* Historical or acute myocardial infarction or ischemia
* Ongoing hypertensive emergency
* Unconsciousness
* Allergic reaction to ketamine
* Increased intracranial or intraocular pressure
* Known pregnancy
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Change in NRS pain scores | Assessed every 6 months.
  The primary outcome measure will be the change in NRS pain scores at ten minutes compared between the subjects administered ketamine and those administered fentanyl.

SECONDARY OUTCOMES:
Rates of adverse events | Assessed every 6 months
  Includes comparisons of clinically significant complications between the two regimens: post-administration respiratory depression as evidenced by either a step up in supplemental oxygen requirements or the need for an airway intervention; episodes of hypotension or hypertension; significant tachycardia; new subjective participant complaints of dysphoria, anxiety, or agitation at any time following drug administration.
Change in NRS pain scores over time | 24 months from start of enrollment
  Evaluate the differences in the slope of the NRS pain scores over time.
Amount of fentanyl required | 24 months from start of enrollment
  Measurement of the total amount of fentanyl/kg body weight/minute of flight that was required to treat patients' pain.
Participant satisfaction | 24 months from start of enrollment
  Overall research participant satisfaction with their level of pain relief at the end of the flight.
Pain Recall | 24 months from start of enrollment
  The subjective ranking of pain recall in comparison to other aspects of the patient's overall episode of care (pre-hospital, emergency department, inpatient, and post-discharge care), as measured at 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Scott T Youngquist, MD, MS, Principal Investigator — University of Utah
Locations (1):
- University of Utah Medical Center, Salt Lake City, Utah, United States